CLINICAL TRIAL: NCT00325754
Title: Benefits of Ambulatory Oxygen in Hypoxemic COPD Patients
Brief Title: Benefits of Lightweight Ambulatory Oxygen Systems for Individuals With Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Chronic Obstructive Pulmonary Disease Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0405S60010; U10HL074424 (NIH); NCT00119860 (obsolete NCT alias)
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E-Cylinder (Active Comparator): 22-lb E-cylinder towed on a cart
  Interventions: Device: E-Cylinder
- Lightweight Cylinder (Active Comparator): 3.6-lb lightweight cylinder that can be carried
  Interventions: Device: Lightweight Cylinder

INTERVENTIONS:
Device: E-Cylinder — Portable Oxygen Therapy Delivered Via An E-Cylinder Mounted On A Wheeled Cart
  Arms: E-Cylinder
Device: Lightweight Cylinder — Ambulatory Oxygen Therapy Delivered Via A Carbon-Wrapped Aluminum Cylinder
  Arms: Lightweight Cylinder

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) affects over 14 million people in the United States. It is the fourth leading cause of death and the only leading cause of death for which mortality rates are rising. Medical science has developed few effective therapies for COPD. In patients with advanced COPD and chronic hypoxemia, long-term oxygen therapy (LTOT) has been shown to be uniquely beneficial. It is the only available non-surgical therapy demonstrated to prolong survival in these patients. This study will compare the clinical and physiologic benefits of two different oxygen therapy devices among hypoxemic individuals with COPD: a lightweight ambulatory oxygen device versus the standard portable E-cylinder device.

DETAILED DESCRIPTION:
Individuals with COPD who experience hypoxemia (reduction of oxygen concentration in arterial blood) have an especially poor prognosis. Provision of LTOT to hypoxemic COPD patients is considered to be the standard of care. The majority of hypoxemic patients that are ambulatory are supplied with pressurized oxygen in E-cylinders. This system weighs approximately 22 pounds, is mounted on a wheeled cart, and is towed by the patient. These cumbersome systems can be seen to impose a significant burden on weak and debilitated patients, discouraging them from being active. E-cylinders towed on a cart are referred to as 'portable', in contrast to lightweight 'ambulatory' oxygen systems, which weigh less than 10 pounds and are designed to be carried by the patient. It is unknown whether patients provided with lightweight ambulatory systems comply better with oxygen prescription and increase their daily level of activity. This study will compare the use and benefits of a lightweight ambulatory oxygen device versus the standard portable E-cylinder device among hypoxemic individuals with COPD. Specifically, the study will examine daily duration of oxygen therapy and activity levels amongst both groups.

ELIGIBILITY:
Inclusion Criteria:

* Currently in a stable phase of COPD, defined as having had no disease exacerbation within the 4 weeks prior to study entry
* Ambulatory
* Forced expiratory volume in one second (FEV1) less than or equal to 60% of predicted value at screening
* Ratio of FEV1 and forced vital capacity (FEV1/FVC) less than or equal to 65% of predicted value at screening
* Currently receiving long-term oxygen therapy (LTOT)
* Partial pressure of oxygen in arterial blood (PaO2) less than 60 torr

Exclusion Criteria:

* Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, left-sided heart failure, peripheral vascular disease, exertional angina, complex arrhythmias, severe dependent edema, ischemic changes on stress electrocardiogram that would be contraindications for unrestricted ambulation or the 6-minute walk test)
* Orthopedic impairments that would limit ambulation
* Participation in the active phase of pulmonary rehabilitation within the 3 months prior to study entry
* Neurologic impairments (e.g., Parkinson's disease or a stroke) or mental states (e.g., senile dementia) that would limit independent ambulation
* Neoplastic disease that is anticipated to influence survival
* Currently receiving lightweight ambulatory oxygen therapy
* Inability to maintain an oxygen saturation of 92% at rest with 4 liter/minute of continuous oxygen flow and during exercise with an oxygen conserver setting of 6 utilizing a nasal cannula
* Currently a smoker
* Sleep apnea if it is characterized primarily as central sleep apnea syndrome (whether being treated or not) OR if it is known or suspected obstructive sleep apnea that has existed for at least 2 months and has not received stable treatment (stable treatment modes include positive airway pressure therapies or dental orthotic/mandibular positioning devices); individuals with diagnosed obstructive sleep apnea must have a body mass index less than or equal to 30 kg/m2 to be eligible for this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K. Albert, Principal Investigator — Denver City-County Health/Hospitals Department; William Bailey, Principal Investigator — University of Alabama at Birmingham; Richard Casaburi, Principal Investigator — Harbor-UCLA Research & Education Institution; John Connett, Principal Investigator — University of Minnesota; Gerard J. Criner, Principal Investigator — Temple University; Stephen C. Lazarus, Principal Investigator — Univeristy of California at San Francisco; Fernando J. Martinez, Principal Investigator — University of Michigan; Dennis E. Niewoehner, Principal Investigator — Minnesota Veterans Medical Research and Education Foundation; John J. Reilly, Principal Investigator — Brigham and Women's Hospital; Steven M. Scharf, Principal Investigator — University of Maryland, College Park; Frank Sciurba, Principal Investigator — University of Pittsburgh
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Francisco, San Francisco, California
  - Harbor-UCLA Research & Education Institution, Torrance, California
  - Denver City-County Health/Hospitals Department, Denver, Colorado
  - University of Maryland Baltimore, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Veterans Research Institute, Minneapolis, Minnesota
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hecht A, Ma S, Porszasz J, Casaburi R; COPD Clinical Research Network. Methodology for using long-term accelerometry monitoring to describe daily activity patterns in COPD. COPD. 2009 Apr;6(2):121-9. doi: 10.1080/15412550902755044. PMID 19378225
- [Result] Casaburi R, Porszasz J, Hecht A, Tiep B, Albert RK, Anthonisen NR, Bailey WC, Connett JE, Cooper JA Jr, Criner GJ, Curtis J, Dransfield M, Lazarus SC, Make B, Martinez FJ, McEvoy C, Niewoehner DE, Reilly JJ, Scanlon P, Scharf SM, Sciurba FC, Woodruff P; COPD Clinical Research Network. Influence of lightweight ambulatory oxygen on oxygen use and activity patterns of COPD patients receiving long-term oxygen therapy. COPD. 2012 Feb;9(1):3-11. doi: 10.3109/15412555.2011.630048. PMID 22292592
- [Derived] Kunisaki KM, Niewoehner DE, Connett JE; COPD Clinical Research Network. Vitamin D levels and risk of acute exacerbations of chronic obstructive pulmonary disease: a prospective cohort study. Am J Respir Crit Care Med. 2012 Feb 1;185(3):286-90. doi: 10.1164/rccm.201109-1644OC. Epub 2011 Nov 10. PMID 22077070

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E-Cylinder | Lightweight Cylinder
Started | 11 | 11
Completed | 7 | 10
Not Completed | 4 | 1
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-Cylinder | Lightweight Cylinder | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.0) | 67.1 (8.1) | 66.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 6 | 8 | 14
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Cigarette Pack Years [Mean (Standard Deviation); unit: pack-years] | 56.5 (31.2) | 50.2 (20.1) | 53.3 (26.0)
Forced expiratory volume in 1 second (FEV1) % Predicted [Mean (Standard Deviation); unit: Percent predicted] | 30.1 (7.7) | 37.1 (13.0) | 31.3 (10.0)
Partial pressure of O2 (PaO2) [Mean (Standard Deviation); unit: torr] | 53.7 (6.0) | 49.5 (6.5) | 51.7 (6.4)
Partial pressure of carbon dioxide (PaCO2) [Mean (Standard Deviation); unit: torr] | 47.5 (7.2) | 45.4 (7.5) | 46.5 (7.3)
Negative logarithm of hydrogen Ion concentration in arterial blood (pHa) [Mean (Standard Deviation); unit: pH units] | 7.42 (0.03) | 7.42 (0.03) | 7.42 (0.03)

OUTCOME MEASURES:

1. Primary Outcome: Stationary Oxygen Use Daily
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | E-Cylinder | Lightweight Cylinder
Number analyzed (Participants) | 7 | 10
Hours | 15.5 (5.5) | 17.0 (4.9)

2. Primary Outcome: Ambulatory/Portable Oxygen Use Daily
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | E-Cylinder | Lightweight Cylinder
Number analyzed (Participants) | 7 | 10
Hours | 1.4 (1.0) | 1.9 (2.4)

3. Primary Outcome: Stationary Oxygen Use Daily
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | E-Cylinder | Lightweight Cylinder
Number analyzed (Participants) | 7 | 10
Hours | 17.6 (4.2) | 16.9 (5.4)

4. Secondary Outcome: Average Mid-day Activity Monitoring at 3 Months
Description: Physical activity was monitored for 3 weeks before the 3-month visit using tri-axial accelerometers worn on a waist belt. Activity is expressed in vector magnitude units (VMU, the vectorial sum of activity counts in three orthogonal directions) per minute. Mid-day defined as 10AM-4PM.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: Vector magnitude units (VMU)/min
Arm/Group | E-Cylinder | Lightweight Cylinder
Number analyzed (Participants) | 11 | 11
Vector magnitude units (VMU)/min | 81.4 (36.0) | 133.6 (75.3)

5. Secondary Outcome: Mid-day Activity Monitoring at 6 Months
Description: Physical activity was monitored for 3 weeks before the 6-month visit using tri-axial accelerometers worn on a waist belt. Activity is expressed in vector magnitude units (VMU, the vectorial sum of activity counts in three orthogonal directions) per minute. Mid-day defined as 10AM-4PM.). Mid-day defined as 10AM-4PM.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Vector magnitude units (VMU)/min
Arm/Group | E-Cylinder | Lightweight Cylinder
Number analyzed (Participants) | 7 | 10
Vector magnitude units (VMU)/min | 90.4 (45.1) | 124.2 (73.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | E-Cylinder | Lightweight Cylinder
Serious Adverse Events (participants affected / at risk) | 5/11 | 4/11
Other Adverse Events (participants affected / at risk) | 8/11 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-Cylinder (N=11) | Lightweight Cylinder (N=11)
Angioedema (Endocrine disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Shortness of Breath (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-Cylinder (N=11) | Lightweight Cylinder (N=11)
Acute Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Other COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Other Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated Blood Urea Nitrogen (BUN) (Renal and urinary disorders) | 0 (0) | 1 (2)
Cystitis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The Data Safety and Monitoring Board requested termination of this study due to low recruitment. 22 participants were randomized out of a goal of 100.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No